CLINICAL TRIAL: NCT00282516
Title: "Internet-based Home Monitoring and Education of Children With Asthma is Comparable to Ideal, Office-based Care: Results of a One-year, Asthma In-Home Monitoring (AIM) Trial"
Brief Title: Asthma In-Home Monitoring (AIM) Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tripler Army Medical Center (U.S. Federal Agency)
Collaborators: U.S. Army Medical Research Acquisition Activity (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 28H01
Record Dates: First submitted 2006-01-25; First posted 2006-01-26 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Mild, Moderate and Severe Persistent Asthma as Defined by NHLBI-2 Guidelines
Keywords: asthma; telemedicine; case management; clinic; children; pediatric
MeSH Terms: conditions — Lymphoma, Follicular; Asthma

INTERVENTIONS:
Procedure: In-home telemonitoring of pediatric patients with persistent asthma

SUMMARY:
OBJECTIVE: Determine whether home asthma telemonitoring using store-and-forward technology improves outcomes when compared to in-person, office-based visits.

DETAILED DESCRIPTION:
OBJECTIVE: Determine whether home asthma telemonitoring using store-and-forward technology improves outcomes when compared to in-person, office-based visits.

METHODS: 120 patients 6-17 yrs with persistent asthma were randomized into two groups: office or virtual. Both groups followed the same ambulatory clinical pathway for 12 months. Office patients received traditional in-person education and case management. Virtual patients received computers, Internet connection, and in-home Web-based case management and received education via the study web site. They also recorded and forwarded a video of peak flow and inhaler use to their case manager two times a week for 6 weeks then once a week thereafter and submitted daily asthma diaries electronically via the web site. Virtual patients were seen in-person only 3 times. Regimen adherence was assessed by monitoring therapeutic (controller medication use, video medication use) and diagnostic (asthma symptom diary and peak flow submitted electronically) outcomes. Disease control outcome measures included quality of life, utilization of services, and symptom control.

RESULTS: 120 volunteers (45 females) were enrolled. The groups were clinically comparable: office 22 females, 38 males 9.0 + 3.0 yrs (mean + SD) virtual 23 females, 37 males, 10.2 + 3.1 yrs. Virtual patients had higher metered-dose inhaler/valved holding chamber score than the office group at 52 weeks (94% vs 89%, p < 0.05), a higher adherence to daily asthma symptom diary submission (35.4% vs 20.8 %, p < 0.01), less participant time (636 vs 713 patient months, p < 0.05), and were older (10.2 + 3.1 years virtual, 9.0 + 3.0 office, p < 0.05). Caregivers in both groups perceived an increase in quality of life (p<0.05) and an increase in asthma knowledge scores from baseline (p < 0.01). There were no other outcome differences in therapeutic or disease control or outcome measures.

CONCLUSION: Virtual patients achieved excellent asthma therapeutic and disease control outcomes. When compared to idealized office-based care they were more adherent to diary submission and had better inhaler scores at 52 weeks than office-based patients. Store-and-forward telemedicine technology and case management provides an additional tool to assist in the management of children with persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of persistent asthma as defined using the NHLBI Expert Panel Report -2 guidelines Assignment of severity classification will be made at the beginning of the study based on severity of disease off therapy.
* Dependent of active duty or retired US military personnel
* 6 to 17 years of age
* Not moving from Oahu for 12 months after entry into study
* Ability to receive cable modem hook-up in home
* Willingness to learn to record and send MDI + spacer technique and peak flow two times week
* Willing to attend asthma education follow-up visits either in person or electronically at 2- weeks, 6- weeks, 3-months and 6-month intervals after initiation into the study.
* Willing to complete survey at the end of study period.
* Willing to sign informed, written consent

Exclusion Criteria:

* Diagnosis of mild intermittent asthma as defined by Expert Panel Report -2 guidelines.
* <6 and >17 years of age
* Family leaving Oahu within 12 months
* Inability to receive cable modem hook-up in home
* Unwilling or unable to learn to record and send MDI + spacer technique and peak flow and/or to attend asthma education follow-up visits either in person or electronically at initiation into study and at 2- weeks, 6- weeks, 3-months and 6 month intervals.
* Unwilling to complete survey at the end of study period.
* Patients or parents who decline to participate.
* Patients with other chronic pulmonary disease (cystic fibrosis, bronchopulmonary dysplasia)

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2003-04; Primary Completion 2004-04 (Actual); Study Completion 2004-04

CONTACTS AND LOCATIONS:
Overall Officials: Charles W Callahan, DO, Principal Investigator — Chief, Department of Pediatrics, Tripler Army Medical Center; Debora S Chan, PharmD, Study Director — Department of Pediatrics, Tripler Army Medical Center
Locations (1):
- Tripler Army Medical Center, Tripler AMC, Hawaii, United States